CLINICAL TRIAL: NCT01397747
Title: Multi-Target Colorectal Cancer Screening Test for the Detection of Colorectal Advanced Adenomatous Polyps and Cancer: DeeP-C Study
Brief Title: Multi-Target Colorectal Cancer Screening Test for the Detection of Colorectal Advanced Adenomatous Polyps and Cancer
Acronym: DeeP-C
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Exact Sciences 2011-01
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Neoplasms; Digestive System Diseases; Colonic Diseases; Colorectal Cancer
Keywords: Cancer; Colorectal Cancer; Neoplasm; Colorectal Neoplasm; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Digestive System Diseases; Colonic Diseases; Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual stool samples may be archived for further research. Clinical data and samples will be kept in a manner that preserves anonymity of the subjects, using the subject ID as the only tracking information. Specimens will be stored in a commercial biorepository contracted by Exact Sciences or at Exact Sciences and may be used for future research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Average risk patients: Subjects will be men and women, 50-84 years of age, inclusive, who are at average risk of developing colorectal cancer.

SUMMARY:
The primary objective is to determine the sensitivity and specificity of the Exact Colorectal Cancer (CRC) screening test for colorectal cancer, using colonoscopy as the reference method. Lesions will be confirmed as malignant by histopathologic examination.

The secondary objective is to compare the performance of the Exact CRC screening test to a commercially available FIT assay, both with respect to cancer and advanced adenoma. Lesions will be confirmed as malignant or precancerous by colonoscopy and histopathologic examination.

DETAILED DESCRIPTION:
Patients who are at average risk of developing colorectal cancer who are eligible for colorectal cancer screening will be asked to collect a single stool sample for the Exact CRC screening test and for the commercially available FIT assay. Subjects will undergo colonoscopy within 90 days of enrollment. Representative histopathology slides from tissue biopsied or excised during colonoscopy and representative histopathology slides resulting from subsequent definitive surgery may be retrieved in order to be evaluated by central pathology to confirm diagnosis and staging.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is average risk for development of colorectal cancer (as defined by the inclusion and exclusion criteria below).
2. Subject is able and willing to undergo a screening colonoscopy within 90 days of enrollment.
3. Subject is 50 to 84 years of age inclusive.
4. Subject is able to comprehend, sign, and date the written informed consent document to participate in the study.
5. Subject is able and willing to provide stool samples according to written instructions provided to them.

Exclusion Criteria:

1. Subject has any condition which, in the opinion of the investigator should preclude participation in the study.
2. Subject has undergone colonoscopy within the previous nine (9) years.
3. Subject has undergone any double-contrast barium enema, virtual (CT-based) colonoscopy, or flexible sigmoidoscopy within the previous five (5) years.
4. Subject has a history of colorectal cancer or adenoma.
5. Subject has a history of aerodigestive tract cancer.
6. Subject has had a positive fecal occult blood test or FIT within the previous six (6) months.
7. Subject has had a prior colorectal resection for any reason other than sigmoid diverticular disease.
8. Subject has had overt rectal bleeding, e.g., hematochezia or melena, within the previous 30 days. (Blood on toilet paper, after wiping, does not constitute rectal bleeding).
9. Subject has a diagnosis or personal history of any of the following high-risk conditions for colorectal cancer:

   * Inflammatory bowel disease (IBD) including chronic ulcerative colitis (CUC) and Crohn's disease.
   * >= 2 first-degree relatives who have been diagnosed with colon cancer. (Note: first-degree relatives include parents, siblings and offspring).
   * One first-degree relative with CRC diagnosed before the age of 60.
   * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP).
   * Hereditary non-polyposis colorectal cancer syndrome (also referred to as "HNPCC" of "Lynch Syndrome").
   * Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Gardner's Syndrome, Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Cronkhite-Canada Syndrome, Neurofibromatosis and Familial Hyperplastic Polyposis.
10. Subject has a family history of:

    * Familial adenomatous polyposis (also referred to as "FAP").
    * Hereditary non-polyposis colorectal cancer syndrome (also referred to as "HNPCC" or "Lynch Syndrome").
11. Participation in any "interventional" clinical study within the previous 30 days in which an experimental treatment is administered or might be administered through a randomized assignment of the subject to one or more study groups.

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at average risk of developing colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 12776 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Imperiale, MD, Principal Investigator — Principal Study Investigator
Locations (174):
- United States (172):
  - Achieve Clinical Research, Birmingham, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Desert Sun Clinical Research, LLC, Tucson, Arizona
  - HealthCare Partners, Alhambra, California
  - HealthCare Partners, Arcadia, California
  - Valley Gastro Consultants, Arcadia, California
  - Desert Oasis Healthcare, Bermuda Dunes, California
  - HealthCare Partners, Burbank, California
  - REMEK Research, Chino, California
  - Southern California Oncology, Downey, California
  - HealthCare Partners Medical Group, El Monte, California
  - Southern California Oncology, Fullerton, California
  - HealthCare Partners, Glendale, California
  - Valley Gastro Consultants, Glendora, California
  - HealthCare Partners, Huntington Park, California
  - Health Care Partners Medical Group, Long Beach, California
  - Health Care Partners San Antonio, Long Beach, California
  - VA Hospital, Long Beach, California
  - Healthcare Partners Medical Group, Los Angeles, California
  - HealthCare Partners, Los Angeles, California
  - Southern California Oncology, Lynwood, California
  - Facey Medical Foundation, Mission Hills, California
  - Healthcare Partners- Mission Plaza, Mission Hills, California
  - Healthcare Partners-Mission Hills, Mission Hills, California
  - REMEK Research, Montclair, California
  - HealthCare Partners Medical Group, Montebello, California
  - Monterey Bay GI Consultants Medical Group & Research Institute, Monterey, California
  - Furtura Research, Monterey Park, California
  - Healthcare Partners Medical Group, Monterey Park, California
  - Diverse Research Solutions, Oxnard, California
  - Desert Oasis Healthcare, Palm Springs, California
  - Desert Regional Medical Center, Palm Springs, California
  - HealthCare Partners, Pasadena, California
  - REMEK Research, Pomona, California
  - Health Care Partners, Redondo Beach, California
  - Institute for Medical Research, Sacramento, California
  - Sharp-Rees-Stealy Medical Group, San Diego, California
  - Sansum Clinic, Santa Barbara, California
  - Santa Monica Research Institute, Santa Monica, California
  - Health Care Partners Medical Group, Torrance, California
  - South Bay Gastroenterology Medical Group, Torrance, California
  - Tujunga Medical Group, Tujunga, California
  - Healthcare Partners-Valencia, Valencia, California
  - Healthcare Partners- Van Nuys, Van Nuys, California
  - Southern California Oncology, Yorba Linda, California
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Gastroenterology Associates of Fairfield County, Fairfield, Connecticut
  - Metropolitan Gastroenterology Group, PC, Washington D.C., District of Columbia
  - Mayo Clinic Florida, Jacksonville, Florida
  - Melbourne GI Center, Melbourne, Florida
  - MIMA Century Research Associates, Melbourne, Florida
  - Suncoast Research Group, Miami, Florida
  - GI Care Center, Miami, Florida
  - Gastro Health P.L., Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Cancer Coalition of South Georgia, Albany, Georgia
  - Phoebe Digestive Health Center, Albany, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Hiram, Georgia
  - Atlanta Gastroenterology Associates, Marietta, Georgia
  - Atlanta Gastroenterology Associates, Woodstock, Georgia
  - NCH Medical Group, Arlington Heights, Illinois
  - Northwest Community Hospital, Arlington Heights, Illinois
  - NCH Medical Group, Buffalo Grove, Illinois
  - Jesse Brown VAMC, Chicago, Illinois
  - Union Health Services, Chicago, Illinois
  - VA Hospital, Hines, Illinois
  - Southwest Gastroenterology, New Lenox, Illinois
  - Union Health Services, Norridge, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Avicenna Clinical Research, Palos Heights, Illinois
  - Rockford Gastroenterology Associates, LTD, Rockford, Illinois
  - Roudebush VA Medical Center, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Gastroenterology & Nutritional Medical Services, Bastrop, Louisiana
  - Gastroenterology Associates, Baton Rouge, Louisiana
  - MGAGI Diagnostic and Therapeutic Center, Metairie, Louisiana
  - New Orleans Research Institute, Metairie, Louisiana
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Digestive Disease Associates, PA, Baltimore, Maryland
  - Gastrointestinal Diagnostic Center, Baltimore, Maryland
  - Metropolitan Gastroenterology Group, Chevy Chase, Maryland
  - Banks Hepatology Institute P.C., College Park, Maryland
  - Digestive Disease Associates, Columbia, Maryland
  - Howard County GIDC, Columbia, Maryland
  - Russell Schub, Columbia, Maryland
  - Columbia Medical Practice, Columbia, Maryland
  - Gasro Center of Maryland, Columbia, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Gastroenterology Associates, Elkridge, Maryland
  - CBM Pathology, Gaithersburg, Maryland
  - Maryland Digestive Disease Center, Laurel, Maryland
  - Gastroenterology Associates, Pasadena, Maryland
  - Boston Medical Center: Center for Digestive Disorders, Boston, Massachusetts
  - Boston Medical Center: Family Medicine, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Shapiro Ambulatory Care Center: Adult Primary Care, Boston, Massachusetts
  - Shapiro Ambulatory Care Center: Women's Health Group, Boston, Massachusetts
  - Commonwealth Clinical Studies PLLC, Brockton, Massachusetts
  - Commonwealth Clinical Studies PLLC, East Bridgewater, Massachusetts
  - Gastrointestinal Specialists, Taunton, Massachusetts
  - Center for Digestive Health, Troy, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Advanced Research Institute, Reno, Nevada
  - Summit Medical Group, Berkeley Heights, New Jersey
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Binghamton Gastroenterology, Binghamton, New York
  - Gastrointestinal Research Group, Great Neck, New York
  - Faculty Practice Associates, New York, New York
  - GI Clinic, New York, New York
  - Internal Medicine Associates, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Practice Associates, New York, New York
  - Digestive Health Specialists, PA, Advance, North Carolina
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - MediSpect, Boone, North Carolina
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - Carolina Digestive Health Associates, Concord, North Carolina
  - Carolina Digestive Health Associates, Davidson, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Carolina Digestive Health Associates, Harrisburg, North Carolina
  - Digestive Health Specialists, PA, Kernersville, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Hanover Medical Specialists, Wilmington, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wilmington Gastroenterology Associates, Wilmington, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Ohio GI & Liver Institute, Cincinnati, Ohio
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Northwest Gastroenterology Clinic, LLC, Portland, Oregon
  - Main Line Gastroenterology, Bala-Cynwyd, Pennsylvania
  - Regional Gastroenterology Associates of Lancaster, Ephrata, Pennsylvania
  - Main Line Gastroenterology, Havertown, Pennsylvania
  - Regional Gastroenterology Associates of Lancaster, Lancaster, Pennsylvania
  - Main Line Gastroenterology, Malvern, Pennsylvania
  - Main Line Gastroenterology, Media, Pennsylvania
  - Main Line Gastroenterology, Perkasie, Pennsylvania
  - PGC Endoscopy Center Inc., Philadelphia, Pennsylvania
  - Main Line Gastroenterology, Wynnewood, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Gastroenterology Associates, Bristol, Tennessee
  - Gastro One, Germantown, Tennessee
  - Gastroenterology Associates of Clinical Research, Kingsport, Tennessee
  - Professional Quality Research, Inc., Austin, Texas
  - Gastroenterology Associates, PA, Houston, Texas
  - Advanced Clinical Research of Houston, Houston, Texas
  - Houston Medical Research Associates, Houston, Texas
  - Professional Quality Research, Inc., Round Rock, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - Advanced Research Institute, Logan, Utah
  - Advanced Research Institute, Ogden, Utah
  - Salt Lake Research, PLLC, Salt Lake City, Utah
  - Advanced Research Institute, Sandy City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Gastroenterology Associates of Tidewater, Norfolk, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Lakeview Medical Center, Suffolk, Virginia
  - Gastroenterology Associates of Tidewater, Virginia Beach, Virginia
  - Northwest Gastroenterology Associates, Bellevue, Washington
  - Marshfield Clinic-Eau Claire Center, Eau Claire, Wisconsin
  - University of Wisconsin Milwaukee, Franklin, Wisconsin
  - UW Health West Clinic, Madison, Wisconsin
  - University of Wisconsin Madison, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - University of Wisconsin Milwaukee, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Clinic-Weston Center, Weston, Wisconsin
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Alberta Health Services, Calgary, Alberta

REFERENCES:
- [Result] Imperiale TF, Ransohoff DF, Itzkowitz SH, Levin TR, Lavin P, Lidgard GP, Ahlquist DA, Berger BM. Multitarget stool DNA testing for colorectal-cancer screening. N Engl J Med. 2014 Apr 3;370(14):1287-97. doi: 10.1056/NEJMoa1311194. Epub 2014 Mar 19. PMID 24645800
- [Derived] Imperiale TF, Gagrat ZD, Krockenberger M, Porter K, Ziegler E, Leduc CM, Matter MB, Olson MC, Limburg PJ. Algorithm Development and Early Performance Evaluation of a Next-Generation Multitarget Stool DNA Screening Test for Colorectal Cancer. Gastro Hep Adv. 2024 May 17;3(6):740-748. doi: 10.1016/j.gastha.2024.05.002. eCollection 2024. PMID 39280922
- [Derived] Ebner DW, Rushlow D, Mou J, Porter K, Finney Rutten LJ, Limburg P, Sancar F, Imperiale TF. Stool-Based Colorectal Cancer Screening Test Performance Characteristics in Those With and Without Hemorrhoids. Mayo Clin Proc Innov Qual Outcomes. 2023 Jul 19;7(4):320-326. doi: 10.1016/j.mayocpiqo.2023.06.003. eCollection 2023 Aug. PMID 37502338

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12,776 participants provided written informed consent. 1,760 could not be evaluated (464- withdrew consent, 1,168- did not undergo colonoscopy, 128- did not submit stool sample).
Groups:
- Average Risk Patients: Subjects will be men and women, 50-84 years of age, inclusive, who are at average risk of developing colorectal cancer. We compared a noninvasive, multitarget stool DNA test with fecal immunochemical test (FIT) in persons at average risk for colorectal cancer. Results were compared to colonoscopy and histopathology was performed on any biopsy or excised lesions.
Period: Overall Study
Arm/Group | Average Risk Patients
Started | 11016
Completed | 9989
Not Completed | 1027
Not completed — Multitarget DNA test excluded | 689
Not completed — Colonoscopy excluded | 304
Not completed — FIT excluded | 34

BASELINE CHARACTERISTICS:
Population: All evaluable participants except for participants who had multitargeted sDNA or colonoscopy excluded.
Arm/Group | Average Risk Patients
Number analyzed (Participants) | 10023
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5378
  Male | 4645
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 991
  Not Hispanic or Latino | 9028
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 36
  Asian | 259
  Native Hawaiian or Other Pacific Islander | 23
  Black or African American | 1071
  White | 8422
  More than one race | 206
  Unknown or Not Reported | 6
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.83 (5.836)
Smoking History [Number; unit: participants]
  Never Smoked | 5531
  Former Smoker | 3589
  Current Smoker | 903

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of the Exact CRC Screening Test With Comparison to Colonoscopy, Both With Respect to Cancer.
Description: An optical colonoscopic procedure is the reference method. Lesions will be confirmed as malignant by histopathologic examination. The DNA test includes quantitative molecular assays for KRAS mutations, aberrant NDRG4 and BMP3 methylation, and Beta-actin, plus a hemoglobin immunoassay. Results were generated with the use of a logistic-regression algorithm, with values of 183 or more considered to be positive. FIT values of more than 100 ng of hemoglobin per milliliter of buffer were considered to be positive. Tests were processed independently of colonoscopic findings. The test functions as a screening tool by generating a score, based on the detection of hemoglobin and multiple DNA methylation and mutational markers, together with an assessment of the total amount of human DNA in each sample. Sensitivity= 100*(multitarget DNA or FIT positive test/positive colonoscopy); Specificity= 100*(multitarget DNA or FIT negative test/negative colonoscopy).
Time Frame: 90 Days
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- Multitarget DNA Test Results: Subjects will be men and women, 50-84 years of age, inclusive, who are at average risk of developing colorectal cancer. We compared a noninvasive, multitarget stool DNA test in persons at average risk for colorectal cancer. Results were compared to colonoscopy and histopathology was performed on any biopsy or excised lesions.
- FIT Test Results: Subjects will be men and women, 50-84 years of age, inclusive, who are at average risk of developing colorectal cancer. We compared a fecal immunochemical test (FIT) in persons at average risk for colorectal cancer. Results were compared to colonoscopy and histopathology was performed on any biopsy or excised lesions.
Arm/Group | Multitarget DNA Test Results | FIT Test Results
Number analyzed (Participants) | 9989 | 9989
percent
  Sensitivity for any Colorectal Cancer | 92.3 [83.0 to 97.5] | 73.8 [61.5 to 84.0]
  Sensitivity Stage I to III | 93.3 [83.8 to 98.2] | 73.3 [60.3 to 83.9]
  Sensitivity CRC and HGD | 83.7 [75.1 to 90.2] | 63.5 [53.5 to 72.7]
  Sensitivity Advanced precancerous lesions | 42.2 [38.9 to 46.0] | 23.8 [20.8 to 27.0]
  Sensitivity nonadvanced adenoma | 17.2 [15.9 to 18.6] | 7.6 [6.7 to 8.6]
  Specificity nonsignificant findings | 86.6 [85.9 to 87.2] | 94.9 [94.4 to 95.3]
  Specificity negative results colonoscopy | 89.8 [88.9 to 90.7] | 96.4 [95.8 to 96.9]

ADVERSE EVENTS:
Description: Only device related adverse events were collected.
Arm/Group | Average Risk Patients
Serious Adverse Events (participants affected / at risk) | 0/11016
Other Adverse Events (participants affected / at risk) | 0/11016

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No